CLINICAL TRIAL: NCT01888588
Title: Risk of Uncomplicated Peptic Ulcer in the General Population
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5040N00006
Record Dates: First submitted 2013-03-18; First posted 2013-06-28 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Peptic Ulcer [Iowa Type (107680.0010)]
Keywords: Uncomplicated peptic ulcer; Low dose aspirin (ASA); Acid-suppressing drugs; Epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients with symptomatic peptic ulcer (UPU)
  Interventions: Drug: Risk of symptomatic peptic ulcer
- Control group: Control group without symptomatic peptic ulcer (UPU).
  Interventions: Drug: Risk of symptomatic peptic ulcer

INTERVENTIONS:
Drug: Risk of symptomatic peptic ulcer — Current use of drugs (ASA; NSAIDs, SSRI,PPI, H2RA) versus non-use

SUMMARY:
The analyses are conducted in a previous population-based cohort study using The Health Improvement Network database in the UK (Cai et al 2009).The aims of the post hoc analyses are:

To estimate the relative risk of uncomplicated symptomatic peptic ulcer (UPU) associated with use of low dose aspirin (ASA) and other anti-inflammatory drugs (NSAIDs, steroids) in the general population To estimate the dose-response and duration-response associated with use of these drugs To estimate the relative risk of UPU associated with naive/non-naive use of low dose ASA in the general population To evaluate the effect of proton pump inhibitors (PPI) (alone or in combination with anti-inflammatory drugs) on the occurrence of UPU in the general population To investigate the management of low dose ASA/oral antiplatelets after UPU

DETAILED DESCRIPTION:
Risk of uncomplicated peptic ulcer in the general population

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 40-84 years in 1997-2005 ( see study population description)

Exclusion Criteria:

- Patients aged below age 40 and 85 years and above ( see study population description)

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is conducted using The Health Improvement Network database in the UK. Patients aged 40-84 years between January 1997 and December 2005 with a registration status of permanent or deceased, who were enrolled for at least 2 years with a GP and had 1 year of electronic prescription history. Patients with a code for cancer, peptic ulcer (both uncomplicated and complicated), upper GI bleeding, oesophageal varices, Mallory-Weiss disease, alcohol abuse, liver disease, or coagulopathies before beginning date were excluded from the source population. All patients in the study population were followed up until the end of the study period (December 2005), or until they reached the age of 85, died, met any of the exclusion criteria (including receiving a diagnosis of complicated peptic ulcer disease), or received a diagnosis of uncomplicated peptic ulcer disease.Patient records were manually reviewed to validate cases.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Relative risk (ratio) of uncomplicated peptic ulcer (UPU) associated with low dose ASA, other antiinflammatory drugs and other common drugs for chronic diseases(paracetamol, SSRI, tricyclic antidepressants, anticoagulants, acid suppressing drugs) | From Januar 1 1997 till December 31 2005, an expected average of 4 years.
  Relative risk (ratio) of UPU associated with current use of the different types of drugs versus non-use.
Management of aspirin after uncomplicated peptic ulcer (UPU). | From January 1, 1997 till december 31, 2005, an average of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Garcia Rodriguez, MD, Principal Investigator — CEIFE (Centro Espanol de Investigacion Farmacoepidemiologica - Spanish Centre for Pharmacoepidemiologic Research )
Locations (1):
- Research Site, Madrid, Spain

REFERENCES:
- [Background] Gonzalez-Perez A, Saez ME, Johansson S, Nagy P, Garcia Rodriguez LA. Risk factors associated with uncomplicated peptic ulcer and changes in medication use after diagnosis. PLoS One. 2014 Jul 8;9(7):e101768. doi: 10.1371/journal.pone.0101768. eCollection 2014. PMID 25003908
- See also: D5040N00006.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=461&filename=D5040N00006.pdf
- See also: D5040N00006_Redacted_Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=461&filename=EPI-Abbreviated_Study_protocol_UPU_gen_pop_D5040N00006_Redacted.pdf